CLINICAL TRIAL: NCT01174498
Title: Controlled, Randomized Study of Pain Perception and Psychophysiological Reactions of the Autonomic Nervous System Under Transcutaneous, Electrical Stimulation of the Vagus Nerve in Healthy Volunteers
Brief Title: Pilot Study of the Effect of Transcutaneous Stimulation of the Vagus Nerve on Pain Perception and Parameters of the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: cerbomed GmbH (Industry)
Responsible Party: Chief Medical Officer, cerbomed GmbH
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: cMPsPAI01
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Pain
Keywords: discomfort; distress; hurt; sting
MeSH Terms: conditions — Pain; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- t-VNS sytem Vagus stimulation (Active Comparator): Subjects experience a transcutaneous vagal stimulation by the t-VNS device
  Interventions: Device: Cerbomed t-VNS® transcutaneous stimulation
- Sham transcutaneous stimulation (Sham Comparator): Sham stimulation with an attached t-VNS device
  Interventions: Device: t-VNS Sham stimulation

INTERVENTIONS:
Device: Cerbomed t-VNS® transcutaneous stimulation — Subjects experience a transcutaneous, electrical, vagal stimulation with the t-VNS device.
  Other Names: Cerbomed t-VNS®
  Arms: t-VNS sytem Vagus stimulation
Device: t-VNS Sham stimulation — t-VNS Sham stimulation
  Arms: Sham transcutaneous stimulation

SUMMARY:
The increased incidence of pain syndromes requires the investigation of pathophysiological coherences as well as searching for new therapies. In the recent years neurostimulating techniques have been a promising approach regarding their analgesic effect. Combined with therapeutic standard procedures they can increase these effects and can have a positive impact on co-morbid diseases. The stimulation of the vagus nerve was proved as an efficient analgesic method in animal experiments and open clinical pilot studies amongst humans. Despite the lack of controlled approaches applying the method against defined pain syndromes, the stimulation of the vagus nerve has shown up as an effective method treating other psychiatric diseases like depression. The processing of stress, which is involved directly and indirectly in the pathogenesis of pain, seems to be susceptible for vagal stimulation. Compared with invasive methods the transcutaneous stimulation offers obvious advantages concerning appliance and occurrence of side effects. There are no studies so far dealing with the neuromodulatory effect on the handling of pain or the clinical therapy of defined (chronic) pain related diseases using the t-VNS system. The study hypothesis implies a change of experiencing pain when applying the t-VNS in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age: Minimum: 18 years Maximum: no limit
* Both Gender
* Normal psychiatric medical history
* Normal neurological report

Exclusion Criteria:

* Psychiatric disease incl. pain-related diseases
* Subject is on medication
* Abuse of drugs or alcohol until 12 weeks before enrollment in the study
* Actual wearing conditions
* Pronounced lack of sleep within the last 2 days of enrollment
* Excessive consumption of alcohol in the last 2 days
* Peripheral neuropathy
* Severe neurological diseases (cerebrovascular diseases, traumatic brain injury, epilepsy, Morbus Parkinson, dementia, systemic neurologic diseases etc.)
* migraine
* carpal tunnel syndrome or other entrapment syndromes
* missing Informed Consent
* Pregnancy
* active implant (like cochlea implant, VNS, pacemaker)
* severe internistic diseases (e.g. arterial hypertension, respiratory failure)
* malignant diseases within the last five years
* severe acute infections (e.g. HIV, hepatitis)
* diseases of the ENT bodysystem: Hearing loss of the left ear which is treated with an hearing instrument, all dermatologic and infectious diseases which affect the area around the pinna and the ear canal
* Other circumstances that in the opinion of the investigator might be an obstacle for enrolling the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
QST- Quantitative Sensory Testing | twice a day, two days in total
  measurement of pain with the qst method before and after the transcutaneous stimulation

SECONDARY OUTCOMES:
Autonomic function measurement | once a day, two days in total
  assessed by skin conductance response (SCL), skin conductance reaction (SCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie der Universität Regensburg, Regensburg, Bavaria, Germany